CLINICAL TRIAL: NCT06134258
Title: Mechanisms of Fasting Induced Reduction in Energy Expenditure - FIRE Trial
Brief Title: Mechanisms of Fasting Induced Reduction in Energy Expenditure
Acronym: FIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EKNZ_2023-01401
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Fasting
Keywords: Thermogenesis
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: randomized, open label, cross-over, monocentric trial in healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting for 24 hours (Other): Fasting for 24 hours
  Interventions: Other: mixed meal test
- Fasting for 12 hours (Other): Fasting for 12 hours
  Interventions: Other: mixed meal test

INTERVENTIONS:
Other: mixed meal test — mixed meal test after fasting

SUMMARY:
Fasting reduces the energy consumption of the human body. The extent of this adaptation varies significantly between different individuals. The aim of this research project is to investigate how this adaptation of the metabolism is regulated by the body. For this purpose, we will first measure how the so-called basal metabolic rate of the body reacts to a short-term fasting of 24 h in a preliminary study. Those subjects with a particularly pronounced and those subjects with an only slightly pronounced reaction of the basal metabolic rate will be invited to the main study.

Here, in random order (24 h fasting vs. 8 h fasting), the following is compared

* how the basal metabolic rate of the body reacts to the reduced energy intake.
* how the energy metabolism increases after a test meal
* what role in particular the thyroid hormones play in this adaptation. In addition, a sample of the subcutaneous adipose tissue is taken in each case and it is examined how the regulation of metabolic processes at the cellular level.

DETAILED DESCRIPTION:
The extent of this adaptation varies significantly between different individuals. The aim of this research project is to investigate how this adaptation of the metabolism is regulated by the body. For this purpose, we will first measure how the so-called basal metabolic rate of the body reacts to a short-term fasting of 24 h in a preliminary study. Those subjects with a particularly pronounced and those subjects with an only slightly pronounced reaction of the basal metabolic rate will be invited to the main study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years
* Body mass index 18.0 to 27.0 kg/m²
* Exclusion Criteria:
* Chronic conditions necessitating medical treatment (e.g., renal failure, hepatic dysfunction, cardiovascular disease, diabetes mellitus),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Hypothyroidism or hyperthyroidism
* Pregnant, breastfeeding and menopausal women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
change of energy expenditure (EE) determined by indirect calorimetry (kcal per 24h) | 60 minutes after ingestion of test meal
  Difference of EE (determined by indirect calorimetry) between baseline and 60 minutes after ingestion of the liquid test meal. Both measurements will be performed after an overnight fasting period.

SECONDARY OUTCOMES:
Level of free thyroxine | after 24 hours and after 12 hours of fasting
  The thyroid hormone (TH) system is an important regulator of EE. We hypothesize that levels of TH are higher in the "spendthrift" than in the "thrifty" group.
Level of free triiodothyronine | after 24 hours and after 12 hours of fasting
  The thyroid hormone (TH) system is an important regulator of EE. We hypothesize that levels of TH are higher in the "spendthrift" than in the "thrifty" group.
Respiratory quotient (RQ) | after 24 hours and after 12 hours of fasting
  We hypothesize that the participants in the "thrifty" group have a lower proportion of fatty acid metabolism and therefore a higher RQ.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Betz, Principal Investigator — University Hospital, Basel, Switzerland; Christian Wolfrum, Study Chair — ETH Zurich
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollstein T, Heinitz S, Basolo A, Krakoff J, Votruba SB, Piaggi P. Reduced metabolic efficiency in sedentary eucaloric conditions predicts greater weight regain in adults with obesity following sustained weight loss. Int J Obes (Lond). 2021 Apr;45(4):840-849. doi: 10.1038/s41366-021-00748-y. Epub 2021 Jan 21. PMID 33479452
- [Background] Reinhardt M, Schlogl M, Bonfiglio S, Votruba SB, Krakoff J, Thearle MS. Lower core body temperature and greater body fat are components of a human thrifty phenotype. Int J Obes (Lond). 2016 May;40(5):754-60. doi: 10.1038/ijo.2015.229. Epub 2015 Oct 26. PMID 26499440
- [Background] Schlogl M, Piaggi P, Pannacciuli N, Bonfiglio SM, Krakoff J, Thearle MS. Energy Expenditure Responses to Fasting and Overfeeding Identify Phenotypes Associated With Weight Change. Diabetes. 2015 Nov;64(11):3680-9. doi: 10.2337/db15-0382. Epub 2015 Jul 16. PMID 26185280
- [Background] Maushart CI, Senn JR, Loeliger RC, Kraenzlin ME, Muller J, Becker AS, Balaz M, Wolfrum C, Burger IA, Betz MJ. Free Thyroxine Levels are Associated with Cold Induced Thermogenesis in Healthy Euthyroid Individuals. Front Endocrinol (Lausanne). 2021 Jun 14;12:666595. doi: 10.3389/fendo.2021.666595. eCollection 2021. PMID 34194392
- [Background] Redman LM, Smith SR, Burton JH, Martin CK, Il'yasova D, Ravussin E. Metabolic Slowing and Reduced Oxidative Damage with Sustained Caloric Restriction Support the Rate of Living and Oxidative Damage Theories of Aging. Cell Metab. 2018 Apr 3;27(4):805-815.e4. doi: 10.1016/j.cmet.2018.02.019. Epub 2018 Mar 22. PMID 29576535
- [Background] Oeckl J, Janovska P, Adamcova K, Bardova K, Brunner S, Dieckmann S, Ecker J, Fromme T, Funda J, Gantert T, Giansanti P, Hidrobo MS, Kuda O, Kuster B, Li Y, Pohl R, Schmitt S, Schweizer S, Zischka H, Zouhar P, Kopecky J, Klingenspor M. Loss of UCP1 function augments recruitment of futile lipid cycling for thermogenesis in murine brown fat. Mol Metab. 2022 Jul;61:101499. doi: 10.1016/j.molmet.2022.101499. Epub 2022 Apr 22. PMID 35470094
- [Background] Pontzer H, Yamada Y, Sagayama H, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SG, Close GL, Cooper JA, Cooper R, Das SK, Dugas LR, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Martin C, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl C, Luke AH, Rood J, Schoeller DA, Westerterp KR, Wong WW, Speakman JR; IAEA DLW Database Consortium. Daily energy expenditure through the human life course. Science. 2021 Aug 13;373(6556):808-812. doi: 10.1126/science.abe5017. PMID 34385400